CLINICAL TRIAL: NCT05779358
Title: The Effects of Bread Consumption on Intestinal and Extra-intestinal Symptoms in Non-coeliac Gluten Sensitivity
Brief Title: Gluten and (Extra-)Intestinal Symptoms in NCGS
Acronym: WoW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Collaborators: University of Leeds (Other); Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NL64850.068.18; METC183011 (Other: Maastricht University)
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Non-celiac Gluten Sensitivity
Keywords: Non-Coeliac Gluten Sensitivity; NCGS; Gluten; Gastrointestinal symptoms
MeSH Terms: interventions — Glutens

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessor know expectancy (E+ or E-) but is blinded to the actual gluten intervention (G+ or G-).
  Participants are told the expectancy, but are unaware of the actual nature of the intervention: they are unaware that there is a 50% chance of receiving either G+ or G- bread, regardless of what they were told.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- E+ G+ (Active Comparator): Participants with the expectation of receiving gluten-containing bread and actually receiving gluten-containing oat bread during the test day.
  Interventions: Other: Expectancy and gluten
- E+ G- (Active Comparator): Participants with the expectation of receiving gluten-containing bread, but actually receiving gluten-free oat bread during the test day.
  Interventions: Other: Expectancy and gluten
- E- G+ (Active Comparator): Participants with the expectation of receiving gluten-free bread but actually receiving gluten-containing oat bread during the test day.
  Interventions: Other: Expectancy and gluten
- E- G- (Placebo Comparator): Participants with the expectation of receiving gluten-free bread and actually receiving gluten-free oat bread during the test day.
  Interventions: Other: Expectancy and gluten

INTERVENTIONS:
Other: Expectancy and gluten — Effect of expectancy to receive gluten and/or actual gluten intake

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled study is to investigate the effect of expectancy related to gluten consumption versus actual gluten intake on overall GI symptoms in individuals with non-coeliac gluten sensitivity (NCGS)

The main questions it aims to answer are:

* what is the effect of consumer expectancy, related to either gluten-containing or gluten-free oat bread, on short-term (within 8 hours) overall GI symptoms in individuals with NCGS?
* what is the effect of actual gluten intake on short-term (within 8 hours) overall GI symptoms in individuals with NCGS

Participants will be randomised into four groups:

1. Participants with the expectation of receiving gluten-containing bread and actually receiving gluten-containing oat bread during the test day. (E+ G+)
2. Participants with the expectation of receiving gluten-containing bread, but actually receiving gluten-free oat bread during the test day. (E+ G-)
3. Participants with the expectation of receiving gluten-free bread but actually receiving gluten-containing oat bread during the test day. (E- G+)
4. Participants with the expectation of receiving gluten-free bread and actually receiving gluten-free oat bread during the test day. (E- G-)

DETAILED DESCRIPTION:
One on-site test, starting with baseline measurement (T = 0). Thereafter, subjects are told that they will receive two slices of gluten-containing bread (E+) or gluten-free bread (E-). Consequently, they receive breakfast with two slices of bread (gluten-containing (G+) or gluten-free (G-)).

After breakfast, questionnaires will be completed every hour for 8 hours. After T = 4 hours, participants receive lunch with two slices of the same bread, combined with the same expectancy, that they received at breakfast.

Follow-up measurements include the same questionnaires at the end of day 1 (from end of test day until they go to sleep), at the end of day 2 and at the end of day 3.

ELIGIBILITY:
Inclusion Criteria:

* Develops self-reported GI symptoms within 8 hours after a single intake of gluten-containing products, without a diagnosis of an organic GI disease;
* Following of willing to follow a gluten-free or gluten-restricting diet (based on a gluten-free dietary compliance questionnaire of Biagi et al. (only group 2, 3 and 4 will be eligible), for at least 1 week prior to study participation and willing to continue with this throughout the study;
* Asymptomatic or only mildly symptomatic (overall (GI) symptom score with VAS < 30mm) while on the gluten-free diet;
* Willing to participate in a study in which they have to consume 4 slices of gluten-containing or gluten-free bread for breakfast and lunch during the test day;
* Willing and able to give written informed consent and to understand, participate and comply with the research project requirements.

Exclusion Criteria:

* Coeliac disease;
* Wheat allergy;
* Presence of an organic GI disease (such as inflammatory bowel disease) or other disease which may interfere with NCGS symptoms (upon judgment of the physician clinical investigator);
* Previous major abdominal surgery or radiotherapy interfering with GI function:

  * Uncomplicated appendectomy, cholecystectomy and hysterectomy allowed unless within the past 6 months;
  * Other surgery may be allowed based upon judgment of the physician-clinical investigator;
* Use of medication potentially influencing GI function and/or NCGS symptoms is allowed, provided that dosing has been stable for > 6 weeks before enrolment;
* Administration of antibiotics, probiotic or prebiotic supplements, investigational drugs or participation in any scientific intervention study, which may interfere with this study (to be decided by the principle investigator), in the 14 days prior to the study
* Excessive use of alcohol (>15 alcoholic units per week), or other drugs;
* Plan to lose weight or follow a specific diet within the study period;
* Any malignancy;
* Pregnancy or breastfeeding;
* Insufficient fluency of the Dutch (for Maastricht and Wageningen) or Englisch (for Leeds) language.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Overall gastrointestinal symptom score (short term) | Test day: baseline (T = 0 hours), hourly after breakfast (T = 1 hour until T = 4 hours), and hourly after lunch (T = 5 hours until T = 8 hours)
  Change from baseline, measured on a Visual Analogue Scale ranged from 0-100, in which 0 is absence of symptoms and 100 is severe symptoms.

SECONDARY OUTCOMES:
Individual gastrointestinal symptom scores (short term) | Test day: baseline (T = 0 hours), hourly after breakfast (T = 1 hour until T = 4 hours), and hourly after lunch (T = 5 hours until T = 8 hours)
  Change from baseline, measured on a Visual Analogue Scale ranged from 0-100, in which 0 is absence of symptoms and 100 is severe symptoms.
  Parameters: abdominal pain, abdominal discomfort, belching, bloating, flatulence, diarrhoea, constipation, urge to empty bowel, fullness, nausea.
Individual extra-intestinal symptom scores (short term) | Test day: baseline (T = 0 hours), hourly after breakfast (T = 1 hour until T = 4 hours), and hourly after lunch (T = 5 hours until T = 8 hours)
  Change from baseline, measured on a Visual Analogue Scale ranged from 0-100, in which 0 is absence of symptoms and 100 is severe symptoms.
  Parameters: tiredness, headache, foggy mind
Average stool frequency and consistency (short term) | Test day: baseline (T = 0 hours), hourly after breakfast (T = 1 hour until T = 4 hours), and hourly after lunch (T = 5 hours until T = 8 hours)
  Bristol Stool Scale, a validated scale for faecal frequency and consistency, by classifying faeces into seven groups. Type 1: separate hard lumps, like nuts (hard to pass); Type 2: sausage-shaped but lumpy; Type 3: Like a sausage but with cracks on its surface; Type 4: Like a sausage or snake, smooth and soft; Type 5: Soft blobs with clear-cut edges (passed easily); Type 6: fluffy pieces with ragged edges, a mushy stool; Type 7: watery, no solid pieces / entirely liquid. Type 1-2 indicate constipation, type 3-4 are ideal stools as they are easier to pass, and type 5-7 may indicate diarrhoea and urgency.
Mood (short term) | Test day: baseline, every hour after breakfast (T = 1 hour until T = 8 hours)
  Change from baseline. Mood is measured by the Positive and Negative Affective Schedule (PANAS) questionnaire.
Overall and individual gastrointestinal symptom score (long-term) | Follow-up: end of day 1 (time from end of test day (t = 8 hours) until end of that day), end of day 2, end of day 3
  Change from baseline, measured on a Visual Analogue Scale ranged from 0-100, in which 0 is absence of symptoms and 100 is severe symptoms.
  Parameters: overall gastrointestinal symtoms, abdominal pain, abdominal discomfort, belching, bloating, flatulence, diarrhoea, constipation, urge to empty bowel, fullness, nausea.
Individual extra-intestinal symptom scores (long term) | Follow-up: end of day 1 (time from end of test day (t = 8 hours) until end of that day), end of day 2, end of day 3
  Change from baseline, measured on a Visual Analogue Scale ranged from 0-100, in which 0 is absence of symptoms and 100 is severe symptoms.
  Parameters: tiredness, headache, foggy mind
Average stool frequency and consistency (long term) | Follow-up: end of day 1 (time from end of test day (t = 8 hours) until end of that day), end of day 2, end of day 3
  Bristol Stool Scale, a validated scale for faecal frequency and consistency, by classifying faeces into seven groups. Type 1: separate hard lumps, like nuts (hard to pass); Type 2: sausage-shaped but lumpy; Type 3: Like a sausage but with cracks on its surface; Type 4: Like a sausage or snake, smooth and soft; Type 5: Soft blobs with clear-cut edges (passed easily); Type 6: fluffy pieces with ragged edges, a mushy stool; Type 7: watery, no solid pieces / entirely liquid. Type 1-2 indicate constipation, type 3-4 are ideal stools as they are easier to pass, and type 5-7 may indicate diarrhoea and urgency.
Mood (long term) | Follow-up: end of day 1 (time from end of test day (t = 8 hours) until end of that day), end of day 2, end of day 3
  Change from baseline. Mood is measured by the Positive and Negative Affective Schedule (PANAS) questionnaire.

OTHER OUTCOMES:
Participant characteristics in relation to NCGS | Data on medical history, demographic factors and adherence to gluten-free diet during the screening visit as part of the screening process. Data on psychological factors will be collected after inclusion of subjects, before the start of the test day.
  To characterise NCGS subjects, data will be collected on medical history (e.g. surgery, GI diseases, medication use, allergies), demographic (e.g. age, gender, educational background, BMI, smoking, alcohol use), adherence to gluten-free diet, and psychosocial factors (relating to e.g. anxiety, depression, somatisation) using screening questionnaires.
Food intake and medication use | Follow-up: end of day 1 (time from end of test day (t = 8 hours) until end of that day), end of day 2, end of day 3
  To check for possible confounders of the follow-up days, a food and medication record will be kept during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Daisy MAE Jonkers, Prof, PhD, Principal Investigator — Maastricht University; Louise Dye, Prof, PhD, Principal Investigator — University of Leeds
Locations (3):
- Netherlands (2):
  - Maastricht University, Maastricht
  - Wageningen University, Wageningen
- University of Leeds, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Graaf MCG, Lawton CL, Croden F, Smolinska A, Winkens B, Hesselink MAM, van Rooy G, Weegels PL, Shewry PR, Houghton LA, Witteman BJM, Keszthelyi D, Brouns FJPH, Dye L, Jonkers DMAE. The effect of expectancy versus actual gluten intake on gastrointestinal and extra-intestinal symptoms in non-coeliac gluten sensitivity: a randomised, double-blind, placebo-controlled, international, multicentre study. Lancet Gastroenterol Hepatol. 2024 Feb;9(2):110-123. doi: 10.1016/S2468-1253(23)00317-5. Epub 2023 Nov 28. PMID 38040019